CLINICAL TRIAL: NCT02831985
Title: Postoperative Controls of Ventilation Tubes in Children - by General Practitioner or Otolaryngologist? A Multicenter Randomized Controlled Trial (The ConVenTu Study)
Brief Title: Postoperative Controls of Ventilation Tubes in Children - by General Practitioner or Otolaryngologist?
Acronym: ConVenTu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Alesund Hospital (Other); Kristiansund Hospital (Other); Molde Hospital (Other); Helse Stavanger HF (Other Government); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ISM-INM/2015/03-1
Record Dates: First submitted 2016-02-19; First posted 2016-07-13 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Otitis
Keywords: Child; Middle ear ventilation; Follow-up studies; General practitioners
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general practice follow-up (Experimental): post-surgery follow-up by general practitioner
  Interventions: Procedure: general practice follow-up
- ENT specialist follow-up (Active Comparator): post-surgery follow-up by ear-nose-throat (ENT) specialist
  Interventions: Procedure: ear-nose-throat (ENT) specialist follow-up

INTERVENTIONS:
Procedure: general practice follow-up — Post-surgery follow-up by general practitioner
  Arms: general practice follow-up
Procedure: ear-nose-throat (ENT) specialist follow-up — Post-surgery follow-up by ear-nose-throat (ENT) specialist
  Arms: ENT specialist follow-up

SUMMARY:
A large number of children with otitis media undergo surgery with ventilation tubes (VTs) placed in the tympanic membrane. This is done to improve hearing and speech development and to reduce ear complaints. The long-term results of VTs are unclear. Follow-up care is required to assure that the tubes are functional, hearing loss has been corrected, and potential complications are properly diagnosed and managed. Guidelines regarding follow-up care give different advices concerning when, how and by whom the controls should be made.

The primary goal of this study is to investigate if follow-up care after surgery with VTs of children aged 3-10 years can be done by general practitioners instead of specialists without negative consequences for the patient.

In the study the child's hearing and speech development, middle ear function, subjective complaints and complications will be assessed. User satisfaction and other aspects related to the quality of control will also be assessed.

If the study shows that follow-ups after surgery with VTs can be done on the level of primary care without loss of care quality, specialist health care services will be spared and cost-effectiveness for the overall healthcare system will improve.

DETAILED DESCRIPTION:
Remark: the change in age range of included children from 4-10 to 3-10 was approved by REK (ethics committee) in November 2018.

ELIGIBILITY:
Inclusion Criteria:

* Insertion of a ventilation tube in at least one ear
* patient at Trondheim University Hospital, Molde Hospital, Aalesund Hospital, Kristiansund Hospital, Stavanger Hospital, Hospital North Norway, or Innlandet Hospital in Gjøvik.

Exclusion Criteria:

* Medical syndromes or other co-existing severe disease that possibly result in increased complication rate after insertion of ventilation tubes, i.e. Downs Syndrome, Cystic Fibrosis, Primary Ciliary Dyskinesia
* Auditory processing disorder (APD)
* Severe neurogenic hearing loss (HL) at least one ear (> 50dB HL in frequencies 0.25 - 4.0 KHz)
* Guardians or children who do not master the Norwegian language

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 322 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
audiogram | 2 years
  pure tone thresholds in decibel (dB) at 0.25-0.5-1-2-4 kHz
audiogram | 4 years
  pure tone thresholds in decibel (dB) at 0.25-0.5-1-2-4 kHz

CONTACTS AND LOCATIONS:
Overall Officials: Wencke Moe Thorstensen, PhD, Principal Investigator — Norwegian University of Science and Technology; Anne S Helvik, PhD, Study Director — Norwegian University of Science and Technology
Locations (6):
- Norway (6):
  - Ålesund Sykehus, Ålesund
  - Sykehuset Innlandet Gjøvik, Gjøvik
  - Kristansund Sykehus, Kristiansund
  - Molde Sykehus, Molde
  - Stavanger Sykehus, Stavanger
  - St Olavs Hospital, ØNH-Avdelingn, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yahiro R, Austad B, Helvik AS, Nilsen AH, Salvesen O, Thorstensen WM. Observation or Otolaryngology Surveillance After Ventilation Tube Insertion in Children: The ConVenTu Noninferiority Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Nov 1;151(11):1063-1070. doi: 10.1001/jamaoto.2025.2880. PMID 41066095
- [Derived] Austad B, Nilsen AH, Helvik AS, Albrektsen G, Nordgard S, Thorstensen WM. Postoperative controls of ventilation tubes in children by general practitioner or otolaryngologist? Study protocol for a multicenter randomized non-inferiority study (The ConVenTu study). Trials. 2020 Nov 23;21(1):950. doi: 10.1186/s13063-020-04849-3. PMID 33228735